CLINICAL TRIAL: NCT01836627
Title: Congenital Muscular Dystrophy (CMD) and the Feasibility of Hyperinsufflation Therapy to Slow Rate of Decline in Lung Volume
Brief Title: A Study to Test Lung Stretch Therapy (Hyperinsufflation) in Children With Collagen VI Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Cure CMD (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIN001CMDwHyperinsufflation; R34HL113390 (NIH)
Record Dates: First submitted 2013-04-12; First posted 2013-04-22 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Congenital Muscular Dystrophy
Keywords: Congenital Muscular Dystrophy; Collagen VI Deficiency; Hyperinsufflation; Cough Assist; LAMA2- Muscular Dystrophy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Hyperinsufflation Therapy (Experimental): Treatment group will have 15 minute hyperinsufflation treatments twice a day for one year.
  Interventions: Other: Hyperinsufflation therapy
- Control (No Intervention): The control group will continue with their current daily care

INTERVENTIONS:
Other: Hyperinsufflation therapy — 15 minutes twice a day of hyperinsufflation with Cough Assist® device
  Arms: Treatment Hyperinsufflation Therapy

SUMMARY:
This research study includes children ages 5 to 20 years old with Collagen Type 6 Congenital Muscular Dystrophy or Laminin α2-related muscular dystrophy (LAMA2-MD). The goal of this study is to measure the effect of breathing exercise to stretch the chest in slowing the loss of breathing function. The breathing stretches are done with a machine called Cough Assist®.

The study is being done at Cincinnati Children's Hospital Medical Center and Children's Hospital of Philadelphia. The study involves traveling to one of these 2 centers for 4 visits over 13 months. The study also includes 3 sets of phone visits called Daily Phone Diaries.

Participants will be "randomized" into one of 2 study groups in a 1:1 ratio. The treatment group will use the Cough Assist® machine twice a day for 15 minutes. The control group will continue with their current daily care. The Cough Assist® is a machine that blows air into the lungs (insufflation) and helps pull air out of the lungs. The investigators will be blowing enough air into the lungs to cause a stretch to the chest. This is called hyperinsufflation.

Study visits will last about 5 to 6 hours and will include medical and quality of life questionnaires and pulmonary function tests to determine lung function and the individualized settings to be prescribed for the Cough Assist®.

DETAILED DESCRIPTION:
Congenital muscular dystrophy (CMD) secondary to collagen VI deficiency and Laminin α2-related muscular dystrophy (LAMA2-MD) are distinct genetic neuromuscular disorders presenting from birth. Respiratory failure is the principal cause of morbidity and mortality from the disease. As CMD has no existing treatment, the majority of affected children develop respiratory failure and require non-invasive ventilation between the first and second decades of life. There is evidence that in muscular dystrophy the progressive decrease in lung volume is disproportionally greater than anticipated for the degree of respiratory muscle weakness. Chest wall stiffness and decreased lung elasticity which collectively diminish compliance of the respiratory system are believed to be important contributors to the disproportionate decrease in lung volume. The investigators' research aims at testing the hypothesis that in subjects with CMD Collagen VI and LAMA2-MD, daily passive stretch of the chest wall through lung hyperinsufflation therapy could slow down the annual rate of decline in lung volume, delay the onset of respiratory failure and improve quality of life.

This is a randomized, controlled, interventional study. The intervention consists of an individualized hyperinsufflation titration protocol. The duration of the active protocol will last 12 months. Because CMD presents a limited subject pool, this study is a partnership with Cincinnati Children's Hospital of Cincinnati (CCHMC) and Children's Hospital of Philadelphia (CHOP) with approximately half of the studies being done at each site. Potential subjects will be identified through Cure CMD international registry and disease specific websites to meet the needed number of subjects.

At Visit 1, subjects will have their baseline assessments, QOL (quality of Life) questionnaires, and pressure titration and hyperinsufflation protocol to determine Peak Insufflation Pressure (PIP). Subjects will be given their randomization assignment into either the Treatment or Control arm. Both groups will have pressure titration and hyperinsufflation protocols for Peak Insufflation Pressure (PIP) at each study visit.

For the Treatment Group, participants at Visit 1 will leave with prescription settings on the Cough Assist® device and they will begin the 12 month interventional period with 15 minute, twice daily hyperinsufflation treatments. Between visits, the Treatment group will mail back the information card (SD card) from the Cough Assist to measure adherence. All visits will be identical for both treatment and control group and will include all the activities from Visit 1 except for randomization.

There will be 3 scheduled phone visits for the Daily Phone Diary (DPD) encounters. The DPD is a phone-based diary that tracks patients and / or caregivers through their activities over the past 24 hours using a cued recall procedure. A set of two DPDs (one weekday and one weekend day) is conducted by phone at each of the 3 assessment points.

The investigators anticipate a significant number of subjects will live greater than 100 miles from the research centers. Travel arrangements will be made by family and paid for by the study through additional funding provided by Cure CMD.

ELIGIBILITY:
Inclusion Criteria:

* 5 years through 20.9 years of age
* for non-ambulatory, subjects, vital capacity ≥30 and ≤ 80% predicted within the past 18 months,
* either gender and we will try to recruit equal numbers of male and female, with vital capacity based on the highest value in past 12 months
* confirmed collagen VI CMD by gene mutation or muscle / skin biopsy OR
* confirmed LAMA2-MD by clinical history and muscle / skin biopsy or by gene mutation that are non-ambulatory and not ventilator dependent.

Exclusion Criteria:

* a major medical condition such as diabetes, renal failure, hepatic failure, cancer, or other known systemic disease or any neuromuscular disorder other than the CMD group
* inability to perform reliable Pulmonary Function Test (PFT)
* tracheostomy
* use of daytime ventilatory support
* PFT values for vital capacity >80 or < 30 %

Patients on positive pressure during sleep or who require cough augmentation will not be excluded.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Difference in rate of decline of lung vital capacity between the two groups | Baseline and app. weeks 17, 34, and 52
  vital capacity (VC)= the volume of gas that can be expelled from the lungs from a position of full inspiration, with no limit to duration of inspiration; equal to inspiratory capacity plus expiratory reserve volume

CONTACTS AND LOCATIONS:
Overall Officials: Raouf S Amin, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (2):
- United States (2):
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania